CLINICAL TRIAL: NCT02687230
Title: Phase 1 Study of 89Zr-DFO-HuMab-5B1 (MVT-2163) With HuMab-5B1 (MVT-5873) in Patients With Pancreatic Cancer or Other CA19-9 Positive Malignancies
Brief Title: Phase 1 Imaging Study of 89Zr-DFO-HuMab-5B1 With HuMab-5B1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech Research & Development, Inc. (Industry)
Collaborators: SciQuus Oncology (Unknown)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MV-0815-CP-001.01
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Carcinoma; Tumors That Express CA19-9
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Subjects receive 3 mg of MVT-2163 without the addition of prior MVT-5873.
  Interventions: Drug: MVT-2163
- Cohort 2 (Experimental): Subjects receive 17 mg of MVT-5873 followed by 3 mg of MVT-2163.
  Interventions: Drug: MVT-2163; Drug: MVT-5873
- Cohort 3 (Experimental): Subjects receive 47 mg of MVT-5873 followed by 3 mg of MVT-2163.
  Interventions: Drug: MVT-2163; Drug: MVT-5873

INTERVENTIONS:
Drug: MVT-2163 — MVT-2163 is administered intravenously as a PET imaging agent
  Other Names: 89Zr-DFO-HuMab-5B1
Drug: MVT-5873 — MVT-5873 is administered intravenously as a non-radioactive blocking agent prior to administration of MVT-2163
  Other Names: HuMab-5B1
  Arms: Cohort 2; Cohort 3

SUMMARY:
Open label, nonrandomized, dose-escalation trial of MVT-2163 and MVT-5873 used in performing PET scans. The study is designed to determine the best time and dose of these agents that result in the best PET image of a tumor. Subjects will be seen on days 1, 2, 4, and 7 for imaging and a clinical assessment. The last study visit is on day 28.

DETAILED DESCRIPTION:
This is an open label, nonrandomized, dose-escalation trial of a fixed dose of MVT-2163 and varying antibody masses of MVT-5873. The study is designed to identify an optimal dose (total antibody mass) and optimal timing, for tumor imaging using PET scanning. This trial will include a dose escalation and an expansion phase. During the dose escalation portion of the study, a determination of the optimal time to perform PET imaging will be made. Following the identification of the "optimal" dose and timing, an 10 additional subjects will be imaged using the best dose and timing.

In each portion of the study subjects will have a screening visit and, no more than 28 days later, those who are eligible for the study will receive MVT-2163. Each cohort will have 3-6 subjects. Subjects in cohort 1 will be administered MVT-2163 alone on day 1. Subjects in cohorts 2 and 3 will receive MVT-5873 on day 1, followed approximately 10 minutes later by MVT-2163. Subjects will return for visits to the clinic on days 2, 4, and 7 for additional imaging and safety assessments. A follow-up visit will occur on day 28.

The study will also evaluate the tissue distribution and pharmacokinetics of MVT-2163 and, based on these data, the study will estimate the radiation dosimetry of MVT-2163. Safety assessments will be performed using ECGs, vital signs measurements, assessments of performance status, and clinical laboratory measurements.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent
* Histologically confirmed, locally-advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) or other malignancies known to express CA19-9 positive malignancies
* At least one lesion by CT or MRI ≥ 2 cm
* ECOG performance status of 0 to 2
* Absolute neutrophil count ≥1.50 x 109/L
* Hemoglobin ≥ 9.0 g/dL (in the absence of red blood cell transfusions in the prior 14 days)
* Platelet count >75,000/ mm3
* AST/SGOT, ALT/SGPT ≤2.5 x ULN, unless liver metastases are clearly present, then ≤5.0 x ULN
* Total bilirubin <1.5x the upper limit of normal unless considered due to Gilbert's syndrome in which case, <3x the upper limit of normal
* Serum creatinine (serum or plasma) ≤ 1.5 x ULN or GFR>50 mL/min
* Serum albumin > 3.0g/dL
* Willingness to participate in collection of pharmacokinetic samples
* Willingness to use adequate contraception throughout study and for a period of 90 days last dose of study drug

Exclusion Criteria:

* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Major surgery other than diagnostic surgery within 28 days
* History of anaphylactic reaction to human, or humanized, antibody
* Other on-going cancer therapy or investigational agents (except MVT-5873 )
* Known history of HIV or Hepatitis C
* Pregnant or currently breast-feeding
* Psychiatric illness/social situations that would interfere with compliance with study requirements
* Significant cardiovascular risk including, but not limited to, recent (within 28 days) coronary stenting or myocardial infarction within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Safety of MVT-2163 alone and in combination with MVT-5873 | About 12 months
  Number of subjects with treatment-related adverse events as assessed by CTCAE v4.0 will be collected and compiled
Peak Plasma Concentration (Cmax) of MVT-2163 alone and in combination with MVT-5873 | About 12 months
  Cmax of MVT-2163
Biodistribution of MVT-2163 alone and in combination with MVT-5873 | About 12 months
  The biodistribution of MVT-2163 will be determined by measuring radiation exposure for key organs and tissues
Dose of MVT-5873 required for optimal tumor visualization when combined with a fixed dose of MVT-2163 | About 12 months
  Three doses of MVT-5873 (0, 17, and 47 mg) will be combined with MVT-2163 in order to determine which dose results in the best PET imaging of tumor
Determine the optimal time interval between MVT-2163 dose administration and tumor PET imaging | About 12 months
  Images will be taken on several days over the first week to determine the optimal day for obtaining PET images
Area under the plasma concentration versus time curve (AUC) of MVT-2163 alone and in combination with MVT-5873 | About 12 months
  AUC of MVT-2163
Half-life (T1/2) of MVT-2163 alone and in combination with MVT-5873 | About 12 months
  Half-life (T1/2) of MVT-2163

SECONDARY OUTCOMES:
The ability of MVT-2163 to detect sites of disease (localized and metastatic) in pancreatic cancer and/or other CA19-9 positive malignancies | About 12 months
  PET scans obtained with MVT-2163 will be compared with conventional imaging (CT/MRI) to determine if MVT-2163 based PET scans are capable of detection tumors seen with conventional methods
Radiation dosimetry estimates using quantitative MVT-2163 biodistribution uptake data | About 12 months
  Bio-distribution data will be used to estimate the radiation exposure of key organs and tissues
MVT-2163 PET imaging results in comparison with varying levels of CA19-9 antigen expression by IHC | About 12 months
  A determination will be made as to the effect of varying levels of CA19-9 antigen expression by tumor IHC on the quality of MVT-2163 PET imaging
MVT-2163 PET imaging results in comparison with circulating CA19-9 levels | About 12 months
  A determination will be made as to the effect of circulating levels of CA19-9 on the quality of MVT-2163 PET imaging
Presence of anti-drug antibodies (ADA) using an MVT-5873 ADA assay | About 12 months
  Subjects will be tested for the development of anti-drug antibodies (ADA) against MVT-5873

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tully KM, Tendler S, Carter LM, Sharma SK, Samuels ZV, Mandleywala K, Korsen JA, Delos Reyes AM, Piersigilli A, Travis WD, Sen T, Pillarsetty N, Poirier JT, Rudin CM, Lewis JS. Radioimmunotherapy Targeting Delta-like Ligand 3 in Small Cell Lung Cancer Exhibits Antitumor Efficacy with Low Toxicity. Clin Cancer Res. 2022 Apr 1;28(7):1391-1401. doi: 10.1158/1078-0432.CCR-21-1533. PMID 35046060